CLINICAL TRIAL: NCT06413186
Title: Examining the Effect of Placenta Delivery Method on Postpartum Pain, Bleeding and Comfort of Women: Randomized Controlled Study
Brief Title: Effect of Placenta Delivery Method on Pain, Bleeding and Comfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Şengül Uluçam, midwife, Student on master degree program at Tarsus University Midwife, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sengul Ulucam
Record Dates: First submitted 2024-04-25; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Placenta Abruptio
Keywords: placenta; labor pain; birt comfort; third stage of labor
MeSH Terms: conditions — Abruptio Placentae; Labor Pain | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: This study is a parallel group, randomized controlled study conducted at the public hospital in Tarsus district of Mersin province. It will consist of primiparas (women who will give birth for the first time) who apply to the delivery room of Tarsus State Hospital. The sample of the research was calculated with the G-Power program. The sample size was calculated as 64 primiparous and 128 primiparous in each group. in total. However, assuming that there will be at least 10% data loss during the research, the study will be carried out with a total of 140 primiparas, 70 primiparas in each group. 70 primiparas who meet the inclusion criteria for the study will be assigned to the experimental group (physiological separation of the placenta using a mixed method), and 70 primiparas will be assigned to the control group (controlled cord traction will be used to deliver the placenta). ) through randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delivery of the placenta by mixed method (Experimental): In this group; As soon as the baby is born, 10 IU oxytocin will be administered IV to the woman.
  The newborn will be placed on the mother's chest for skin-to-skin contact, Uterine tone will be evaluated while the baby is at the mother's breast, The cord will be clamped late (after the pulse in the cord stops/within 1-3 minutes after the baby is born), The placenta will be delivered physiologically.
  Interventions: Drug: Uteratonic administration; Other: cord clamping; Other: delivery of the placenta
- Delivery of the placenta by active method (Active Comparator): In this group; As soon as the baby is born, 10 IU oxytocin will be administered IV to the woman.
  The newborn will be placed on the mother's chest for skin-to-skin contact, Uterine tone will be evaluated while the baby is at the mother's breast, The cord will be clamped late (after the pulse in the cord stops/within 1-3 minutes after the baby is born), The placenta will be removed with controlled cord traction.
  Interventions: Drug: Uteratonic administration; Other: cord clamping; Other: delivery of the placenta

INTERVENTIONS:
Drug: Uteratonic administration — Administer IV 10 IU oxytocin
  Other Names: Oxytocin administration
Other: cord clamping — delayed cord clamping
Other: delivery of the placenta — Applying controlled core traction

SUMMARY:
The aim of this thesis is to examine the effect of the placenta delivery method on women's postpartum pain, bleeding and comfort. It is a randomized controlled experimental study. The research will be conducted at Mersin Tarsus state hospital between March 2024 and August 2024. The study will be conducted with 140 primiparous women, 70 primiparous pregnant women in the experimental group and 70 primiparous pregnant women in the control group, who meet the research criteria and apply to the delivery room of Tarsus State Hospital between these dates. The research will be carried out with a control group (those receiving routine hospital protocol/where the placenta is delivered with controlled cord traction) and an experimental group (physiological separation of the placenta with a mixed method). Interventions applied to research groups vary depending on the characteristics of the group. In both groups, interventions in the delivery room will be performed by the researcher midwife. If any complications develop during the research, independent of the interventions, if the woman undergoes a cesarean section, or if situations that meet the exclusion criteria occur, that woman will be excluded from the sample. The researcher will apply a routine hospital birth management protocol to both groups during the first three stages of labor. However, the way the placenta is delivered in the third stage (physiological with mixed management or controlled cord traction with active management) will differ. The researcher will apply the Visual Analogue Scale (VAS) twice, at the beginning and at the end of the third phase of labor, apply the Postpartum Comfort Scale at the 4th postpartum hour, and record hemoglobin and hematocrit values at admission to the hospital, which is the hospital's routine protocol, and in the hemogram test at the 6th hour postpartum. HB and HCT values will be used to interpret the amount of postpartum bleeding. The hypotheses of the research are as follows; H1: In the active management of the 3rd stage of labor, delivery of the placenta with controlled cord traction affects the woman's perception of postpartum pain.

H2: In the active management of the 3rd stage of labor, delivering the placenta with controlled cord traction affects the woman's amount of postpartum bleeding.

H3: In the active management of the 3rd stage of labor, delivering the placenta with controlled cord traction affects the woman's postpartum comfort level.

H4: In the mixed management of the 3rd stage of labor, physiological delivery of the placenta affects the woman's perception of postpartum pain.

H5: In the mixed management of the 3rd stage of labor, physiological delivery of the placenta affects the amount of postpartum bleeding of the woman.

H6: In the mixed management of the 3rd stage of labor, physiological delivery of the placenta affects the woman's postpartum comfort level.

ELIGIBILITY:
Inclusion Criteria:

Agreeing to participate in the research

* No communication problems
* Between 19-35 years old
* 38-42 weeks of gestation
* Having a single and healthy fetus and newborn
* Having a vaginal birth
* Firstborn
* Women who are not at risk during birth and postpartum period

Exclusion Criteria:

Women who develop complications during birth and the postpartum period (placenta not separating, part of the placenta remaining in the uterus, development of atony, manual rupture of the uterus, cord rupture, etc.)

* Those receiving anticoagulant treatment during pregnancy
* The duration of the 3rd stage of labor lasts more than 30 minutes
* Instrumental (using vacuum/forceps) birth

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Skala (VAS) | 15-30 minutes
  It is a scale in which the person marks the part expressing his/her pain on a 10 cm ruler where painlessness and unbearable pain are shown at each end. VAS was preferred because it is easy to use, sensitive in measuring pain intensity, and reliable. In the evaluation of VAS, 0-2 cm indicates "no pain", 3-4 cm indicates "mild pain", 5-6 cm indicates "Moderate pain", 7-8 cm indicates "Severe pain" and 9-10 cm indicates "Unbearable". shows "pain"

SECONDARY OUTCOMES:
Postpartum Comfort Scale | 15-30 minutes
  It was developed by Karakaplan and Yıldız in 2010 to measure the physical, psychospiritual and sociocultural comfort of women giving birth. The scale has a 5-point Likert structure ("totally agree: 5 points" and "strongly disagree: 1 point") and consists of a total of 34 items. "Totally agree" in the positive items in the scale indicates high comfort (5 points), while negative items indicate low comfort (1 point). score). As the scores obtained from the scale increase, it shows that the comfort level increases. As a result of the study, scores close to 170 indicate that the person's comfort is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus üniversitesi, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Begley CM, Guilliland K, Dixon L, Reilly M, Keegan C. Irish and New Zealand midwives' expertise in expectant management of the third stage of labour: the 'MEET' study. Midwifery. 2012 Dec;28(6):733-9. doi: 10.1016/j.midw.2011.08.008. Epub 2011 Oct 19. PMID 22015217
- [Background] Begley CM, Gyte GM, Devane D, McGuire W, Weeks A, Biesty LM. Active versus expectant management for women in the third stage of labour. Cochrane Database Syst Rev. 2019 Feb 13;2(2):CD007412. doi: 10.1002/14651858.CD007412.pub5. PMID 30754073
- [Background] Dixon L, Tracy SK, Guilliland K, Fletcher L, Hendry C, Pairman S. Outcomes of physiological and active third stage labour care amongst women in New Zealand. Midwifery. 2013 Jan;29(1):67-74. doi: 10.1016/j.midw.2011.11.003. Epub 2011 Dec 20. PMID 22188999
- [Background] Herman A, Zimerman A, Arieli S, Tovbin Y, Bezer M, Bukovsky I, Panski M. Down-up sequential separation of the placenta. Ultrasound Obstet Gynecol. 2002 Mar;19(3):278-81. doi: 10.1046/j.1469-0705.2002.00557.x. PMID 11896951
- [Background] Hofmeyr GJ, Mshweshwe NT, Gulmezoglu AM. Controlled cord traction for the third stage of labour. Cochrane Database Syst Rev. 2015 Jan 29;1(1):CD008020. doi: 10.1002/14651858.CD008020.pub2. PMID 25631379
- [Background] Munoz M, Stensballe J, Ducloy-Bouthors AS, Bonnet MP, De Robertis E, Fornet I, Goffinet F, Hofer S, Holzgreve W, Manrique S, Nizard J, Christory F, Samama CM, Hardy JF. Patient blood management in obstetrics: prevention and treatment of postpartum haemorrhage. A NATA consensus statement. Blood Transfus. 2019 Mar;17(2):112-136. doi: 10.2450/2019.0245-18. Epub 2019 Feb 6. PMID 30865585
- [Background] Prendiville WJ, Elbourne D, McDonald S. Active versus expectant management in the third stage of labour. Cochrane Database Syst Rev. 2000;(3):CD000007. doi: 10.1002/14651858.CD000007. PMID 10908457
- [Background] Winter C, Macfarlane A, Deneux-Tharaux C, Zhang WH, Alexander S, Brocklehurst P, Bouvier-Colle MH, Prendiville W, Cararach V, van Roosmalen J, Berbik I, Klein M, Ayres-de-Campos D, Erkkola R, Chiechi LM, Langhoff-Roos J, Stray-Pedersen B, Troeger C. Variations in policies for management of the third stage of labour and the immediate management of postpartum haemorrhage in Europe. BJOG. 2007 Jul;114(7):845-54. doi: 10.1111/j.1471-0528.2007.01377.x. PMID 17567419
- [Background] Gulmezoglu AM, Widmer M, Merialdi M, Qureshi Z, Piaggio G, Elbourne D, Abdel-Aleem H, Carroli G, Hofmeyr GJ, Lumbiganon P, Derman R, Okong P, Goudar S, Festin M, Althabe F, Armbruster D. Active management of the third stage of labour without controlled cord traction: a randomized non-inferiority controlled trial. Reprod Health. 2009 Jan 21;6:2. doi: 10.1186/1742-4755-6-2. PMID 19154621
- [Background] Gunaydin B. Management of Postpartum Haemorrhage. Turk J Anaesthesiol Reanim. 2022 Dec;50(6):396-402. doi: 10.5152/TJAR.2022.21438. PMID 36511487
- [Background] Labor S, Maguire S. The Pain of Labour. Rev Pain. 2008 Dec;2(2):15-9. doi: 10.1177/204946370800200205. PMID 26526404
- [Background] Lowe NK. The nature of labor pain. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S16-24. doi: 10.1067/mob.2002.121427. PMID 12011870
- [Background] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Background] Rabe H, Diaz-Rossello JL, Duley L, Dowswell T. Effect of timing of umbilical cord clamping and other strategies to influence placental transfusion at preterm birth on maternal and infant outcomes. Cochrane Database Syst Rev. 2012 Aug 15;(8):CD003248. doi: 10.1002/14651858.CD003248.pub3. PMID 22895933
- See also: Ekşi Z. (2019). Doğum Sonu Dönem. Hemşirelik ve Ebelik İçin Kadın Sağlığı ve Hastalıkları, Bölüm 12, Arslan Ö.E. (editör), Akademisyen Kitabevi, Ankara. — https://dergipark.org.tr/tr/download/issue-full-file/62207
- See also: Erdemir F, Çırlak A. (2013). Rahatlık kavramı ve hemşirelik kullanımı. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 6(4), 224-230. — https://dergipark.org.tr/tr/download/article-file/753452
- See also: FIGO/ICM Joint Statement. Management of the Third Stage of Labour to Prevent Post-partum Haemorrhage. 2007. — https://www.figo.org/joint-statement-recommendation-uterotonics-prevention-pph
- See also: Güngör İ, Yıldırım-Rathfisch G. (2009). Normal doğum eyleminin ikinci ve üçüncü evresinde kanıta dayalı uygulamalar. Hemşirelikte Araştırma Geliştirme Dergisi, 2:56-65. — https://dergipark.org.tr/tr/download/article-file/984224
- See also: Karakaplan S, Yıldız H.( 2010). Doğum sonu konfor ölçeği geliştirme çalışması. Maltepe Üniversitesi Hemşirelik Bilim ve Sanatı Dergisi, 3(1), 55-65. — https://toad.halileksi.net/olcek/dogum-sonu-konfor-olcegi/
- See also: Kolcaba K. (2003). Comfort theory and practice: a vision for holistic health care and research. Springer Publishing Co, New York — https://books.google.com.tr/books?id=nduGie_ouQkC&pg=PR3&hl=tr&source=gbs_selected_pages&cad=1#v=onepage&q&f=false
- See also: National Institute for Health and Care Excellence. Intrapartum care for healthy women and babies. Intrapartum Care for Healthy Women and Babies, Guideline CG190. London: National Institute for Health and Care Excellence, 2014. — https://www.nice.org.uk/guidance/cg190
- See also: Potur DÇ, Merih YD, Külek H, Gürkan ÖC. (2015). Doğum konforu ölçeğinin Türkçe geçerlik ve güvenirlik çalışması. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 18(4), 252-258. — https://dergipark.org.tr/tr/download/article-file/773243
- See also: Sarı E, Fışkın G, Karakaş S. (2020). Ebelik Öğrencilerinin Doğum Ağrısı ve Yönetimi Hakkındaki Bilgi Düzeylerinin Belirlenmesi. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 23(1), 1-8. — https://dergipark.org.tr/tr/download/article-file/1013476
- See also: T.C. Sağlık Bakanlığı Halk Sağlığı Genel Müdürlüğü Kadın ve Üreme Sağlığı Dairesi Başkanlığı, Doğum Sonu Bakım Yönetim Rehberi, Ankara, 2018. — https://hsgm.saglik.gov.tr/depo/birimler/kadin-ve-ureme-sagligi-db/Rehberler/dogum_sonu_bakim_2020.pdf
- See also: TÜİK (2018). Anne Ölüm Oranı — https://data.tuik.gov.tr
- See also: Türk Neonatoloji Derneği (TND). (2021). Doğum Salonu Yönetimi Rehberi 2021 Güncellemesi. https://www.neonatology. org.tr/wp-content/uploads/2021/08/Dogum-Salonu-Yonetimi- Reh-beri-2021-Guncellemesi-1.pdf — https://neonatology.org.tr/uploads/content/tan%C4%B1-tedavi/6_min.pdf
- See also: Ünal E, Şenol DK (2022). Primipar annelerde doğum şeklinin doğum sonu konfor ve emzirme başarısına etkisi. Ordu Üniversitesi Hemşirelik Çalışmaları Dergisi, 5(2), 158-165. — https://dergipark.org.tr/tr/download/article-file/1654977
- See also: Ünal İ, Can HÖ, Oran NT. (2019). Doğum Eyleminde Ebelik Gereksinimlerinin Orem Özbakım Yetersizlik Kuramına Göre Değerlendirilmesi. Life Sciences, 14(2), 41-47. — https://dergipark.org.tr/tr/download/article-file/708480
- See also: World Health Organization. (2012). WHO recommendations for the prevention and treatment of postpartum haemorrhage. — https://iris.who.int/bitstream/handle/10665/75411/9789241548502_eng.pdf;jsessionid=FF2B57F78B26844C943223EF5CD9E357?sequence=%201
- See also: World Health Organization(2014).Guideline:Delayed umbilical cord clamping for improved maternal and infant health and nutrition outcomes. Geneva: World Health Organization — https://www.who.int/publications/i/item/9789241508209
- See also: Yücel ŞÇ. (2011). Kolcaba'nın Konfor Kuramı. Ege Üniversitesi Hemşirelik Yüksek Okulu Dergisi 27 (2), 79-88. — https://dergipark.org.tr/tr/download/article-file/825497